CLINICAL TRIAL: NCT06790602
Title: A Single-arm, Open-label, Phase II Trial of Cemiplimab Plus Gemcitabine as Second-line Treatment in Patients With Metastatic Pancreatic Adenocarcinoma Harboring SWItch/Sucrose Non-Fermentable (SWI/SNF) Alterations.
Brief Title: Cemiplimab Plus Gemcitabine in Patients With Metastatic Pancreatic Adenocarcinoma
Acronym: SWITCH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Gregory Botta, Associate Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 810575
Record Dates: First submitted 2025-01-16; First posted 2025-01-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma (mPDAC)
Keywords: cemiplimab; gemcitabine; immune checkpoint inhibitors; pancreatic ductal adenocarcinoma; SWI/SNF; combination therapy; PDAC; Phase 2; metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cemiplimab; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Study participants will be treated with intravenous cemiplimab 3mg/kg every 2 weeks and intravenous gemcitabine 1000mg/m^2 on days 1, 8,15 of every 28-day cycle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cemiplimab Plus Gemcitabine (Experimental): Combination therapy of cemiplimab plus gemcitabine. Cemiplimab will be supplied as 350 mg vials for intravenous administration at 3 mg/Kg every 2 weeks. Gemcitabine will be administered intravenously per standard of care at 1000mg/m^2 on days 1, 8, 15 of every 28-day cycle. Cemiplimab plus gemcitabine will be administered until disease progression or other reasons that warrant discontinuation.
  Interventions: Drug: Cemiplimab Plus Gemcitabine

INTERVENTIONS:
Drug: Cemiplimab Plus Gemcitabine — Cemiplimab Plus Gemcitabine
  Other Names: Cemiplimab; Libtayo; REGN2810; Gemzar

SUMMARY:
This is a Phase 2 trial evaluating the combination of cemiplimab with the standard of care chemotherapy agent gemcitabine for the treatment of patients with metastatic pancreatic ductal adenocarcinoma with SWItch/Sucrose Non-Fermentable (SWI/SNF) alterations who have already been treated with FOLFIRINOX (5-fluoruracil, leucovorin, irinotecan, oxaliplatin) or gemcitabine/nab-paclitaxel chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy with FOLFIRINOX (5-fluoruracil, leucovorin, irinotecan, oxaliplatin) or gemcitabine/nab-paclitaxel is the backbone of modern therapy of metastatic pancreatic ductal adenocarcinoma. Generally, the chemotherapy regimen is chosen based on the patient's performance status and ability to tolerate the specific side effect profiles of the two regimens. As many patients with metastatic pancreatic ductal adenocarcinoma suffer from multiple co-morbidities that develop with the disease, they are often subjected to treatment interruptions, dose reductions, and palliative single-agent therapies. Thus, better treatments are needed for this disease. A treatment modality for many cancer types is represented by immune checkpoint inhibitors. However, over 98% of pancreatic ductal adenocarcinoma are deemed 'cold', which means that they have an uninflamed tumor microenvironment incapable of spurring an immune response during therapy with immune checkpoint inhibitors. In fact, immune checkpoint inhibitors such as ipilimumab (Cytotoxic T-lymphocyte Associated protein 4 blocker) and nivolumab (Programmed Cell Death 1 blocker) have not shown efficacy in pancreatic ductal adenocarcinoma as single agents.

Alterations in the chromatin remodeling complex SWI/SNF appear to sensitize tumors to immune checkpoint inhibitors and may be a surrogate biomarker of efficacy of these compounds. In retrospective studies, immune checkpoint inhibitors in SWI/SNF altered pancreatic ductal adenocarcinoma resulted in improved tumor responses and longer progression-free survival and overall survival. In addition, preclinical studies of immune checkpoint inhibitors plus gemcitabine show superior antitumor effects compared to gemcitabine alone in both orthotopic murine pancreatic cancer cell line grafts and in genetically engineered mouse models.

Thus, the investigators propose a clinical trial of the immune checkpoint inhibitor cemiplimab plus standard of care gemcitabine to evaluate efficacy and safety of this combination in patients with metastatic pancreatic ductal adenocarcinoma harboring SWI/SNF alterations who did not respond or were intolerant to the standard of care chemotherapies (FOLFIRINOX or gemcitabine/nab-paclitaxel). The investigators hypothesize that the combination cemiplimab plus gemcitabine will lead to better overall survival, progression free survival, and overall response rate compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Ability to understand the nature of this study, comply with study and follow-up procedures, and give written informed consent.
3. Histologically or cytologically confirmed pancreatic ductal adenocarcinoma. Primary tumor can be intact or post-resection with newly developed metastatic disease.
4. Stage IV disease (measurable disease by Immunotherapeutics Response Evaluation Criteria in Solid Tumors is required).
5. Alterations in SWI/SNF complex chromatin remodeling genes (ARID1A, ARID1B, PBRM1, SMARCA4 and SMARCB1, etc.) detected by next generation sequencing performed prior to enrollment on an ultrasound-guided core biopsy of the primary tumor.
6. One previous line of therapy for pancreatic ductal adenocarcinoma (NOT immunotherapy or cellular therapy).
7. Last dose of chemotherapy administered > 14 days prior to the initiation of study therapy.
8. Last dose of radiation therapy or administered > 28 days prior to the initiation of study therapy.
9. Eastern Cooperative Oncology Group performance score of 0-1.
10. Adequate bone marrow function: Absolute neutrophil count ≥ 1,500 cells per microliter; Platelet count ≥ 100,000 cells per microliter; Hemoglobin ≥ 9.0 grams per deciliter.
11. Adequate hepatic function: Total bilirubin ≤ 1.5 times upper limit of normal (NOTE high bilirubin levels due to Gilbert's syndrome are allowed); Aspartate transaminase ≤ 3.0 times upper limit of normal (≤5.0 times upper limit of normal if liver metastases are present); Alanine transaminase ≤ 3.0 times upper limit of normal (≤5.0 times upper limit of normal if liver metastases are present).
12. Adequate renal function: Serum creatinine ≤ 1.5 times upper limit of normal.
13. Calculated corrected QT Interval (QTcF) average of the triplicate electrocardiograms <470 milliseconds.
14. Participants not of child-bearing potential, or participants of child-bearing potential who agree to use adequate contraceptive measures during the study and for at least 6 months after the last cemiplimab dose; who are not breastfeeding, and who have a negative serum or urine pregnancy test within 72 hours prior to initiation of study therapy.
15. For participants able to cause a pregnancy: use of condoms or other methods to ensure effective contraception with partner during study participation and for at least 6 months after the last cemiplimab dose.

Exclusion Criteria:

1. Two or more lines of systemic or previous investigational therapy for metastatic pancreatic ductal adenocarcinoma.
2. History of any autoimmune disease requiring treatment within the past 12 months prior to enrollment.
3. History of transplanted organ/bone marrow.
4. History of interstitial lung disease.
5. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
6. History of previous malignancy (except in-situ cancer or basal or squamous cell skin cancer) within past 3 years prior to enrollment.
7. History of immune checkpoint inhibitor therapy, ever.
8. Known bleeding disorders (e.g., van Willebrand's disease or hemophilia).
9. Current use of warfarin or other vitamin K antagonists. NOTE: if therapeutic anticoagulation is necessary, low molecular weight heparin or oral factor Xa inhibitors are the anticoagulants of choice.
10. Current use of a strong cytochrome P450 3A inhibitor (for example, antifungal medications, grapefruit juice, amiodarone, etc.).
11. Presence of known central nervous system or brain metastases.
12. History of other diseases, metabolic dysfunction, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that, in the opinion of the investigator, renders the subject at high risk from treatment complications or might affect the interpretation of the results of the study.
13. Life expectancy of <3 months.
14. Known active, not-controlled human immunodeficiency virus, hepatitis B or hepatitis C infection or diagnosis of immunodeficiency.
15. Receipt of a live vaccine within 4 weeks of start of study medication.
16. Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to enrollment.
17. Major surgery within 4 weeks of the start of study treatment. Major surgeries are defined as those surgeries that require general anesthesia. Insertion of a vascular access device, biliary drainage tube, gastrointestinal stent are NOT considered major surgery.
18. Pregnancy or lactation.
19. Known allergic reactions to components of the study intervention, cemiplimab and/or gemcitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 7 months
  To evaluate the overall survival of participants with metastatic pancreatic adenocarcinoma harboring SWI/SNF alterations treated with cemiplimab in combination with gemcitabine as a second-line treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P Botta, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available.

REFERENCES:
- [Background] Botta GP, Kato S, Patel H, Fanta P, Lee S, Okamura R, Kurzrock R. SWI/SNF complex alterations as a biomarker of immunotherapy efficacy in pancreatic cancer. JCI Insight. 2021 Sep 22;6(18):e150453. doi: 10.1172/jci.insight.150453. PMID 34375311